CLINICAL TRIAL: NCT00442611
Title: A Pilot Study to Evaluate the Safety and Efficacy of Abatacept in Patients With Systemic Sclerosis
Brief Title: A Study to Evaluate the Safety and Efficacy of Abatacept in Patients With Diffuse Systemic Sclerosis (Scleroderma)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Lorinda S Chung, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 100 186
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-09

CONDITIONS: Scleroderma, Diffuse; Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Abatacept (Experimental): Abatacept (dosed based upon weight) administered intravenously (IV) on days 1, 15, 30 and monthly thereafter for a total of 7 doses.
  Interventions: Drug: Abatacept
- IV fluid (Placebo Comparator): Placebo to match abatacept (IV fluid) administered on days 1, 15, 30 and monthly thereafter for a total of 7 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept
  Arms: Abatacept
Drug: Placebo
  Arms: IV fluid

SUMMARY:
Systemic sclerosis (scleroderma) is an autoimmune connective tissue disease that involves the skin and other internal organs for which there are few effective treatment options. We hypothesize that treatment with abatacept, a new therapy recently approved for the treatment of rheumatoid arthritis, may reduce the progression of skin thickening and fibrosis in people with scleroderma.

DETAILED DESCRIPTION:
Systemic sclerosis is an autoimmune connective tissue disease of unknown etiology characterized by progressive fibrosis of the skin and internal organs, vascular damage, and autoantibody production. Although the disease is relatively rare, it is associated with considerable morbidity and mortality. There have been improvements in survival over the past few decades; however, this has been related to better management of vascular manifestations of disease including renal crisis, pulmonary hypertension, gastroesophageal reflux disease, and Raynaud's phenomenon. Clinical studies of disease modifying therapies for cutaneous disease to date have been relatively unsuccessful.

Although the etiology of the disease remains unknown, several observations support the role of activated T cells in both the blood and skin of affected patients. Abatacept, a recombinant fusion protein that blocks T cell activation, has recently been approved by the FDA for rheumatoid arthritis. We hypothesize that inhibition of T cell activation with abatacept may be efficacious in the treatment of patients with diffuse systemic sclerosis. This is a randomized, double-blinded, placebo-controlled clinical trial of abatacept versus placebo in patients with diffuse systemic sclerosis. Changes in validated measures of skin thickness and disease activity over 6-months of treatment will be compared between patients receiving abatacept and those receiving placebo. Patients will be randomized 2:1 to receive abatacept.

The protocol was amended during the study and the outcome measures "Change in Serum Autoantibody Profile" and "Change in Serum Cytokine Profile" were changed to exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diffuse systemic sclerosis
* age 18 years or older
* Adequate renal, pulmonary, and cardiovascular function
* Willingness to use effective contraception for the duration of the study if subject is of childbearing potential

Exclusion Criteria:

* Other connective tissues diseases or overlap syndromes including MCTD, SLE, RA, eosinophilic fasciitis, and limited systemic sclerosis or morphea
* Use of disease modifying agents including methotrexate, cyclosporine,azathioprine, mycophenolate mofetil, minocycline, doxycycline, minocycline, thalidomide, penicillamine, tamoxifen, colchicine, or investigational agent within 90 days of screening visit
* HIV, Hepatitis B or Hepatitis C infection
* use of prednisone greater than 10mg daily for 28 days prior to screening visit
* women who are breastfeeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Farmer Chakravarty, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Chakravarty EF, Martyanov V, Fiorentino D, Wood TA, Haddon DJ, Jarrell JA, Utz PJ, Genovese MC, Whitfield ML, Chung L. Gene expression changes reflect clinical response in a placebo-controlled randomized trial of abatacept in patients with diffuse cutaneous systemic sclerosis. Arthritis Res Ther. 2015 Jun 13;17(1):159. doi: 10.1186/s13075-015-0669-3. PMID 26071192

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abatacept | IV Fluid
Started | 7 | 3
Completed | 6 | 3
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept | IV Fluid | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.4) | 48.6 (13.9) | 44.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Rodnan Skin Score
Description: Modified Rodnan Skin Score measures skin thickness and is the sum of scores from 17 surface anatomic areas rated on a 0-3 scale (0=normal skin; 1=mild thickness; 2=moderate thickness; 3=severe thickness with inability to pinch the skin into a fold). Total modified Rodnan Skin Score ranges from 0 (best possible outcome) to 51 (worst possible outcome).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: MRSS score
Arm/Group | Abatacept | IV Fluid
Number analyzed (Participants) | 7 | 3
MRSS score | -8.6 (7.5) | -2.3 (15)

2. Secondary Outcome: Oral Aperture at Baseline and Month 6
Time Frame: Baseline; Month 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Abatacept | IV Fluid
Number analyzed (Participants) | 7 | 3
mm
  Right side baseline | 31.1 (6.51) | 21.0 (4.32)
  Right side month 6 | 29.4 (4.98) | 21.0 (1.41)
  Left side baseline | 30.9 (7.18) | 20.0 (2.45)
  Left side month 6 | 29.3 (4.65) | 20.0 (4.08)

3. Secondary Outcome: Hand Extension at Baseline and Month 6
Time Frame: Baseline; Month 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Abatacept | IV Fluid
Number analyzed (Participants) | 7 | 3
mm
  Right hand baseline | 177.7 (28.11) | 98.3 (20.95)
  Right hand month 6 | 178.9 (31.38) | 103.3 (24.94)
  Left hand baseline | 183.7 (23.96) | 110.7 (35.98)
  Left hand month 6 | 184.3 (25.23) | 116.3 (40.58)

4. Secondary Outcome: Digital Ulcerations at Baseline and Month 6
Time Frame: Baseline; Month 6
Measure: Mean (Standard Deviation); unit: ulcers
Arm/Group | Abatacept | IV Fluid
Number analyzed (Participants) | 7 | 3
ulcers
  Right hand baseline | 0.3 (0.70) | 0.7 (0.47)
  Right hand month 6 | 0.1 (0.35) | 1.3 (0.47)
  Left hand baseline | 0.0 (0.00) | 0.7 (0.47)
  Left hand month 6 | 0.0 (0.00) | 1.0 (0.82)

5. Secondary Outcome: Change in Pulmonary Function Tests
Description: FVC (Forced Vital Capacity) is the amount of air that can be forcibly exhaled from the lungs after taking the deepest possible breath. DLCO (Diffusing capacity of the lung for carbon monoxide) is the extent to which oxygen passes from the lungs to the blood.
Time Frame: 6 months
Population: Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: % Predicted
Arm/Group | Abatacept | IV Fluid
Number analyzed (Participants) | 6 | 3
% Predicted
  FVC % Predicted | 1.3 (8.5) | .3 (8.5)
  DLCO % Predicted | 2.0 (6.3) | -7.4 (10.7)

6. Secondary Outcome: Change in Scleroderma Health Assessment Questionnaire
Description: The HAQ Disability Index (HAQ-DI) includes 20 items in 8 functional domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities) assessing the patient's usual abilities in the past seven days. Each item is scored on a 0-3 scale (0=without any difficulty; 1=with some difficulty; 2=with much difficulty; 3=unable to do). The use of assistive devices for any domain increases the domain score by 1 point to a maximum of 3. The overall score is calculated by summing the highest item score in each of the domains and dividing the sum by 8, with an overall score of 0 indicating no disability, and a score of 3 indicating severe disability.
  The time points compared were 6 months to baseline (6 months minus baseline).
Time Frame: 6 months
Population: Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: HAQ-DI score
Arm/Group | Abatacept | IV Fluid
Number analyzed (Participants) | 6 | 3
HAQ-DI score | -0.04 (.24) | .25 (.25)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Abatacept | IV Fluid
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/3
Other Adverse Events (participants affected / at risk) | 6/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=7) | IV Fluid (N=3)
Infection (Vascular disorders) | 1 (1) | 0 (0) — Infected toe digital ulcer
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Abatacept (N=7) | IV Fluid (N=3)
infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
lower extremity edema (Vascular disorders) | 0 (0) | 1 (1)
headache (General disorders) | 1 (1) | 0 (0)
dry mouth (General disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0/1 (0) | 1 (1)
fever (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No